CLINICAL TRIAL: NCT00273416
Title: A Randomized Double Blind, Placebo Controlled Balanced 4-Way Crossover Study To Assess The Efficacy Of Single Oral Doses Of PF-00592379 On Erectile Function, Using 100mg Sildenafil As A Positive Control
Brief Title: A Randomized Double Blind, Placebo Controlled Balanced 4-Way Crossover Study To Assess The Efficacy Of Single Oral Doses
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A7771002
Record Dates: First submitted 2006-01-04; First posted 2006-01-09 (Estimated); Last update posted 2006-08-24 (Estimated); Status verified 2006-08

CONDITIONS: Impotence
MeSH Terms: conditions — Erectile Dysfunction | interventions — Sildenafil Citrate

INTERVENTIONS:
Drug: PF-00592379
Drug: Sildenafil 100mg

SUMMARY:
The primary aim of this study is to assess how effective PF-00592379 is in restoring penile erections in patients with erectile dysfunction. Patients will attend for 4 treatment visits where they will receive the following in random order; 2 separate doses of PF-00592379, sildenafil 100mg used as a positive control, or placebo (dummy medication). The effect on penile erections will be assessed in the clinic using penile plethysmography (RigiScan PlusTM technique).

ELIGIBILITY:
Inclusion Criteria:

* Erectile dysfunction, previous good response to an oral treatment for erectile dysfunction.

Exclusion Criteria:

* Patients with high blood pressure or certain heart conditions (e.g. angina, heart failure), regardless of whether treated or not.
* Patients on nitrates or alpha-blocker medications.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32
Dates: Start 2006-01

PRIMARY OUTCOMES:
Duration of penile erections of greater than or equal to 60% rigidity as assessed by penile plethysmography (RigiScan PlusTM).

SECONDARY OUTCOMES:
Duration and quality of penile erections recorded in a self-assessment diary.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Pfizer Investigational Site, Oslo, Norway
- Pfizer Investigational Site, Belfast, Northern Ireland, United Kingdom

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7771002&StudyName=A+Randomized+Double+Blind%2C+Placebo+Controlled+Balanced+4%2DWay+Crossover+Study+To+Assess+The+Efficacy+Of+Single+Oral+Doses